CLINICAL TRIAL: NCT03263026
Title: A Randomized Phase 3 Study to Evaluate the Efficacy and Safety of Enzastaurin Plus R-CHOP Versus R-CHOP in Treatment-Naive Subjects With High-Risk Diffuse Large B-Cell Lymphoma Who Possess the Novel Genomic Biomarker DGM1™
Brief Title: Study to Assess Enzastaurin + R-CHOP in Subjects With DLBCL With the Genomic Biomarker DGM1™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DB102-02
Record Dates: First submitted 2017-08-18; First posted 2017-08-28 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma; Non-Hodgkin's Lymphoma; enzastaurin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Following screening (within 28 days), subjects will receive up to 6 cycles of R-CHOP immunochemotherapy (21-day cycles) plus study drug, during the combination phase.
  Combination Phase (6 x 21-day cycles with R-CHOP): Subjects will receive a loading dose of 1125 mg (3 tablets TID) followed by 500 mg (4 tablets QD) of study drug (enzastaurin/placebo) daily.
  Sigle-Agent Phase: Following completion of up to 6 cycles of R-CHOP, subjects in the enzastaurin arm who have a CR, or PR (at investigator's discretion) may continue to take single-agent study drug (enzastaurin 500 mg) daily for up to 2 additional years.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Denovo Biopharma, the study Sponsor, will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- R-CHOP + enzastaurin (Active Comparator): Subjects in the R-CHOP + enzastaurin Arm will receive R-CHOP (Rituximab-375 mg/m2 i.v., Cyclophosphamide-750 mg/m2 i.v., Doxorubicin-50 mg/m2 i.v., Vincristine-1.4 mg/m2 i.v. (2 mg max), and Prednisone-100 mg p.o.), as directed, plus a 1125 mg loading dose of enzastaurin on Day 2 followed by 500 mg daily.
  After completion of the combination phase of treatment, subjects will be reassessed using PET-CT and subsequently each subject's treatment assignment will be unblinded. Subjects randomized to the enzastaurin arm who have CR or PR at investigator's discretion by the Lugano Classification will be offered single-agent enzastaurin at 500 mg/day (4 tablets once daily) continuously for up to 2 additional years. All other subjects on the enzastaurin arm will receive no further study treatment and transition into the follow up phase of the study; these subjects will receive standard of care based on their response assessment.
  Interventions: Drug: Enzastaurin Hydrochloride
- R-CHOP + placebo (Placebo Comparator): Subjects in the R-CHOP + placebo Arm will receive R-CHOP (Rituximab-375 mg/m2 i.v., Cyclophosphamide-750 mg/m2 i.v., Doxorubicin-50 mg/m2 i.v., Vincristine-1.4 mg/m2 i.v. (2 mg max), and Prednisone-100 mg p.o.), as directed, plus an identical number of tablets as the subjects in the enzastaurin Arm.
  After completion of the combination phase of treatment, subjects will be reassessed using PET-CT and subsequently each subject's treatment assignment will be unblinded. All subjects randomized to the placebo arm will receive no further study treatment and transition into the follow up phase of the study; these subjects will receive standard of care based on their response assessment.
  Interventions: Other: R-CHOP + placebo

INTERVENTIONS:
Drug: Enzastaurin Hydrochloride — R-CHOP + Enzastaurin (Kinenza®) 125 mg
  Other Names: Kinenza®
  Arms: R-CHOP + enzastaurin
Other: R-CHOP + placebo — R-CHOP + placebo
  Other Names: Placebo
  Arms: R-CHOP + placebo

SUMMARY:
This randomized, placebo-controlled phase 3 study planned to enroll approximately 235 treatment-naïve subjects with high-risk Diffuse Large B-Cell Lymphoma (DLBCL). Subjects were randomized 1:1 to R-CHOP plus enzastaurin or R-CHOP (plus placebo during induction). All subjects received up to 6 cycles (3 weeks per cycle) of treatment. PET/ CT was used to assess radiographic response at the end of treatment. Each subject's treatment assignment was unblinded after combination phase tumor response assessment. Subjects randomized to the enzastaurin arm who have a complete response (CR) or partial response (PR) (at investigator's discretion) by Lugano Classification had the opportunity to continue in the single-agent phase of the study and receive single-agent enzastaurin for up to 2 additional years.

DETAILED DESCRIPTION:
Diffuse Large B-Cell Lymphoma (DLBCL) is the most common of the Non-Hodgkin's Lymphomas, accounting for between 30%-40% of all cases. The incidence of DLBCL generally increases with age and roughly half of all patients are over the age of 60 at the time of diagnosis.

DLBCL is classified as an aggressive lymphoma meaning that its clinical course can progress rapidly to death. Nevertheless, patients with DLBCL can be cured with the appropriate treatment. The current standard of care treatment for DLBCL consists of rituximab added to the anthracycline-containing combination chemotherapy regimen of cyclophosphamide, doxorubicin, vincristine and prednisone (NCCN Treatment Guidelines). This regimen is referred to as R-CHOP immunochemotherapy. For DLBCL as a whole, R-CHOP immunochemotherapy has resulted in cure rates of approximately 60%. However, for individual patients 5-year survival rates can range from 90% for low-risk patients to less than 50% for high-risk patients.

Most important, for those subjects refractory to R-CHOP therapy less than 10% achieve a durable remission with secondary therapy. Thus, while R-CHOP remains the standard treatment for high-risk, advanced-stage DLBCL, approximately 30-40% of patients fail front-line therapy with most not achieving complete response or with early relapse. An essential step to move forward and improve the outcomes of these patients is to increase the rate of complete response to front-line R-CHOP therapy.

For this reason, there has been a great deal of effort placed on attempting to define disease characteristics that predispose patients to a poorer prognosis with R-CHOP therapy. Molecular and gene expression profiling of tumors and a variety of clinical prognostic indices have been used to identify patients at higher risk of failing R-CHOP immunochemotherapy. While this work has identified subgroups of patients who do not respond well to R-CHOP, to date these efforts have not resulted in substantial gains in response to front-line therapy.

Denovo Biopharma (Denovo) has pioneered an alternative approach to this challenging problem. Denovo has developed a model that employs sophisticated pharmacogenomic testing to detect somatic biomarkers that identify those subjects who responded to a particular study treatment with the aim of re-studying the drug of interest, in this case enzastaurin, in an enriched population.

Applying this technology to archived DNA samples from completed studies of enzastaurin in subjects with DLBCL, Denovo has identified a somatic biomarker that reliably identified subjects for whom the study treatment significantly prolonged survival. Enzastaurin is an oral serine/threonine kinase inhibitor, that targets the PKC, and phosphoinositide 3-kinase (PI3K) and AKT pathways to inhibit tumor cell proliferation, induce tumor cell apoptosis, and suppress tumor-induced angiogenesis.

The purpose of the current study is to prospectively assess the effect on survival of adding enzastaurin to R-CHOP immunochemotherapy in the front-line treatment of an enriched population of subjects with DLBCL.

Enzastaurin, an acyclic bisindolylmaleimide, is a potent and selective inhibitor of PKC-beta. At plasma concentrations achieved clinically, enzastaurin and its metabolites suppress signaling not only through PKC, but also through the PI3K/AKT pathway; these pathways promote tumor-induced angiogenesis, as well as tumor cell survival and proliferation. Accordingly, inhibition of signaling pathways by enzastaurin suppresses the phosphorylation of glycogen synthase kinase 3 beta (GSK3-beta) at ser9, induces cell death (apoptosis), and suppresses proliferation in cultured cell lines from human colon cancers, glioblastoma and lymphomas. Oral dosing with enzastaurin to achieve exposure levels similar to that in human clinical studies suppresses vascular endothelial growth factor (VEGF)-induced angiogenesis and the growth of human colon cancer and glioblastoma xenografts. These studies have demonstrated that enzastaurin can suppress tumor growth through multiple mechanisms: the direct effect of inducing tumor cell death, suppressing tumor cell proliferation, and the indirect effect of suppressing tumor-induced angiogenesis.

ELIGIBILITY:
Inclusion Criteria

1. Male or female at least 18 years of age and able to provide informed consent.
2. Histologically confirmed diagnosis of CD20-positive DLBCL based on the WHO classification (2016); the diagnosis must be confirmed at the enrolling site. Subjects with high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements and high-grade B-cell lymphoma, NOS are eligible.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
4. International Prognostic Index (IPI) score of at least 3.
5. Estimated life expectancy of at least 12 weeks.
6. Adequate organ function as follows (within 14 days prior to randomization):

   1. Hepatic: total bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 5 times ULN in the case of Gilberts Syndrome, liver or pancreatic involvement by lymphoma); alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 times ULN (≤ 5 times ULN if liver involvement)
   2. Renal: creatinine clearance of ≥ 40 mL/min by Cockcroft- Gault equation
   3. Bone marrow: platelets ≥75 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, hemoglobin ≥8 g/dL. (Platelets ≥50 x 109/L, ANC ≥ 1.0 x 109/L, hemoglobin ≥ 7 g/dL permitted if documented bone marrow involvement)
7. Male or female with reproductive potential, must be willing to use an approved contraceptive method (for example, intrauterine device (IUD), birth control pills, or barrier device) during and for 3 months after discontinuation of study treatment. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization.

   1. Men are considered of reproductive potential unless they have undergone a vasectomy and confirmed sterile by a post-vasectomy semen analysis.
   2. Women are considered of reproductive potential unless they have undergone hysterectomy and/or surgical sterilization (at least 6 weeks following a bilateral oophorectomy, bilateral tubal ligation, or bilateral tubal occlusive procedure that has been confirmed in accordance with the device's label) or achieved postmenopausal status (defined as cessation of regular menses for greater than 12 consecutive months in women at least 45 years of age).
8. Left ventricular ejection fraction ≥50% by echocardiography or nuclear medicine multi-gated scan.
9. Must be able to swallow tablets.
10. Must be able to comply with study protocol procedures.
11. Willing to consent to have blood stored for possible future biomarker and disease analysis.
12. Must have available and willing to submit pre-systemic treatment DLBCL tumor biopsy tissue/slides for central pathology review.

Exclusion Criteria

1. Received treatment with an investigational drug within the last 30 days.
2. Receiving or has received radiation or any other systemic anticancer treatment for lymphoma (Up to 7 days of corticosteroids are permitted but must be administered after eligibility IPI determination and imaging scans).
3. History of indolent lymphoma or follicular Grade 3b lymphoma.
4. Primary mediastinal (thymic) large B-cell lymphoma.
5. B-cell lymphoma, unclassifiable, with features. intermediate between DLBCL and classical Hodgkin lymphoma.
6. Burkitt lymphoma.
7. Pregnancy or breastfeeding.
8. Known central nervous system (CNS) involvement.
9. Any significant concomitant disorder based on the discretion of the investigator, including but not limited to active bacterial, fungal, or viral infection, incompatible with participation in the study.
10. A second primary malignancy (except adequately treated non-melanoma skin cancer); subjects who have had another malignancy in the past, but have been disease-free for more than 5 years, and subjects who have had a localized malignancy treated with curative intent and disease free for more than 2 years are eligible.
11. Use of a strong inducer or moderate or strong inhibitor of CYP3A4 within 7 days prior to start of study therapy or expected requirement for use on study therapy.
12. Personal or immediate family history of long QT syndrome, QTc interval >450 msec (males) or >470 msec (females) at screening (recommended that QTc be calculated using Fridericia correction formula, QTcF: see Section 6.2.1), or a history of unexplained syncope.
13. Use of any medication that can prolong the QT/QTc interval within 7 days prior to start of study therapy or expected requirement for use on study therapy.
14. History of severe allergic or anaphylactic reaction to monoclonal antibody therapy.
15. Confirmed diagnosis of progressive multifocal leukoencephalopathy.
16. Ongoing grade 2 or higher peripheral neuropathy.
17. Have any of the following cardiac disorders: uncontrolled hypertension, unstable angina, myocardial infarction within 8 weeks of randomization, New York Heart Association (NYHA) Grade 2 or higher congestive heart failure, ventricular arrhythmia requiring medication within 1 year of randomization, Fontaine Classification stage III or higher peripheral arterial disease.
18. Received a live vaccine within 28 days of study Day 1.
19. HIV positive.
20. Evidence of chronic hepatitis C infection as indicated by antibody to HCV with positive HCV-RNA.
21. Evidence of chronic hepatitis B infection as indicated by either:

    1. HBsAg+ or
    2. HBcAb+ with HBV-DNA+ (any detectable amount is considered positive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (27):
  - Oncology Specialties: Clearview Cancer Institute, Huntsville, Alabama
  - University of Arizona, Tucson, Arizona
  - Central Arkansas Radiation Therapy Institute, Little Rock, Arkansas
  - Desert Hematology, Rancho Mirage, California
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - Norton Cancer Institute Oncology Practices - St. Matthews Location, Louisville, Kentucky
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Mercy Research, Springfield, Missouri
  - Saint Louis University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Norris Cotton Cancer Center Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Summit Medical Group, Morristown, New Jersey
  - Atlantic Health System/ Morristown Meeical Center, Morristown, New Jersey
  - New York Medical College, Hawthorne, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Hematology & Oncology Associates, Inc., Canton, Ohio
  - Tri-County Hematology & Oncology Associates, Inc., Massillon, Ohio
  - Toledo Clinic Cancer Centers, Toledo, Ohio
  - University of Texas Southwestern Medical Center - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Oncology Consultants: Memorial City, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Center Alliance, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Vince Lombardi Cancer Center (Aurora St. Luke's Medical Center), Milwaukee, Wisconsin
- China (12):
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital (Hematology Dept), Beijing
  - JiLin Cancer Hospital（Lymphoma hematology Dept), Changchun
  - West China Hospital of Sichuan University (Hematology Dept), Chengdu
  - Second Affiliated Hospital of Dalian Medical University, Dalian
  - GuangDong General Hospital, Guangzhou
  - ZheJiang Cancer Hospital ( Lymphoma Dept), Hangzhou
  - Harbin Medical University Cancer Hospital (Oncology Internal), Harbin
  - Fudan University Shanghai Cancer Hospital, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - HeNan Cancer Hospital (Hematology Dept), Zhengzhou
  - The First Affiliated Hospital of ZhengZhou University (Oncology Dept), Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nowakowski GS, Zhu J, Zhang Q, Brody J, Sun X, Maly J, Song Y, Rizvi S, Song Y, Lansigan F, Jing H, Cao J, Lue JK, Luo W, Zhang L, Li L, Han I, Sun J, Jivani M, Liu Y, Heineman T, Smith SD. ENGINE: a Phase III randomized placebo controlled study of enzastaurin/R-CHOP as frontline therapy in high-risk diffuse large B-cell lymphoma patients with the genomic biomarker DGM1. Future Oncol. 2020 May;16(15):991-999. doi: 10.2217/fon-2020-0176. Epub 2020 Apr 6. PMID 32250167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intent to treat (ITT) population 254 (126 in R-CHOP plus enzastaurin arm and 128 in R-CHOP plus placebo arm). The DGM1 status was not available for two subjects as these subjects either withdrew consent or died prior to sample collection. Total 256 patients were initially randomized but two patients were not dosed.
Groups:
- R-CHOP + Enzastaurin; R-CHOP + Placebo: The Phase 2 study of enzastaurin used "standard" International Prognostic Index, and therefore the same index will be used in the current study. This index defines 5 variables: age (> 60), tumor stage (III or IV), number of extranodal sites (> 1), ECOG performance status (> 1) and serum lactate dehydrogenase (LDH) (> 1 times upper limit of normal). One point is assigned for each variable and subjects with 3 points are classified as high-intermediate risk, and subjects with 4 or 5 points are classified as high-risk DLBCL. Subjects must have at least 3 points in order to be eligible for this study.
Period: Overall Study
Arm/Group | R-CHOP + Enzastaurin | R-CHOP + Placebo
Started | 128 | 128
Completed | 85 | 99
Not Completed | 43 | 29
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0
Not completed — Other/ Various | 41 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R-CHOP + Enzastaurin | R-CHOP + Placebo | Total
Number analyzed (Participants) | 126 | 128 | 254
Age, Continuous [Median (Full Range); unit: years] | 63 [27 to 86] | 65 [28 to 91] | 65 [27 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 57 | 120
  Male | 63 | 71 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 88 | 89 | 177
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 39 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
DGM1 positive Biomarker status [Count of Participants; unit: Participants] — Population: Two hundred and fifty-six (256) subjects were enrolled in the study (126 in the treatment group and 128 in the placebo group, including 112 and 121 subjects who had the DGM1 biomarker in each group respectively). The DGM1 status was not available for two subjects as these subjects either withdrew consent or died prior to sample collection, therefore not included in ITT (number analyzed).
  Participants | 112 | 121 | 233

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Subjects Who Possess the DGM1™ Biomarker
Description: The primary objective of this study is to compare the effect of R-CHOP/enzastaurin versus R-CHOP alone on overall survival in treatment naive, high-risk subjects with DLBCL who possess the DGM1™ biomarker.
Time Frame: Primary Outcome evaluated at 12 months.
Measure: Number; unit: percentage of patients
Groups:
- RCHOP + Placebo: The Phase 2 study of enzastaurin used "standard" International Prognostic Index, and therefore the same index will be used in the current study. This index defines 5 variables: age (> 60), tumor stage (III or IV), number of extranodal sites (> 1), ECOG performance status (> 1) and serum lactate dehydrogenase (LDH) (> 1 times upper limit of normal). One point is assigned for each variable and subjects with 3 points are classified as high-intermediate risk, and subjects with 4 or 5 points are classified as high-risk DLBCL. Subjects must have at least 3 points in order to be eligible for this study.
Arm/Group | R-CHOP + Enzastaurin | RCHOP + Placebo
Number analyzed (Participants) | 112 | 121
percentage of patients | 82 | 87

2. Secondary Outcome: To Determine the Effect on Overall Survivor of Adding Enzastaurin to R-CHOP in Treatment naïve Subjects With High-risk DLBCL Regardless of DGM1 Biomarker Status.
Description: The secondary outcome of this study is to determine the effect on OS of adding enzastaurin to R-CHOP in treatment naïve subjects with high-risk DLBCL regardless of DGM1 biomarker status.
Time Frame: Secondary Outcome evaluated at 12 months.
Measure: Count of Participants; unit: Participants
Groups:
- R-CHOP + Enzastaurin Hydrochloride: Subjects in the R-CHOP + enzastaurin Arm will receive R-CHOP (Rituximab-375 mg/m2 i.v., Cyclophosphamide-750 mg/m2 i.v., Doxorubicin-50 mg/m2 i.v., Vincristine-1.4 mg/m2 i.v. (2 mg max), and Prednisone-100 mg p.o.), as directed, plus a 1125 mg loading dose of enzastaurin on Day 2 followed by 500 mg daily.
  Enzastaurin Hydrochloride: R-CHOP + Enzastaurin (Kinenza®) 125 mg
- R-CHOP + Placebo: Subjects in the R-CHOP + placebo Arm will receive R-CHOP (Rituximab-375 mg/m2 i.v., Cyclophosphamide-750 mg/m2 i.v., Doxorubicin-50 mg/m2 i.v., Vincristine-1.4 mg/m2 i.v. (2 mg max), and Prednisone-100 mg p.o.), as directed, plus an identical number of tablets as the subjects in the enzastaurin Arm.
  R-CHOP + placebo: R-CHOP + placebo
Arm/Group | R-CHOP + Enzastaurin Hydrochloride | R-CHOP + Placebo
Number analyzed (Participants) | 126 | 128
Participants | 100 | 100

3. Other Pre Specified Outcome: Presence of Chromaturia as a Predictor of Efficacy
Description: Urine color will be analyzed by the central lab and overall survival will be determined for subjects with reddish discoloration of the urine. Testing may be performed to define the chemical profile of the urine.
Time Frame: 3.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from enrollment till the end of the study participation or death, whichever comes first, up to 42 months.
Arm/Group | R-CHOP + Enzastaurin | R-CHOP + Placebo
All-Cause Mortality (participants affected / at risk) | 68/126 | 77/128
Serious Adverse Events (participants affected / at risk) | 75/126 | 59/128
Other Adverse Events (participants affected / at risk) | 126/126 | 125/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP + Enzastaurin (N=126) | R-CHOP + Placebo (N=128)
(Product Issues) | 75 | 59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP + Enzastaurin (N=126) | R-CHOP + Placebo (N=128)
WBC Decreased (Investigations) | 85 | 72
Neutrophil Count Decreased (Investigations) | 80 | 81
Platelet Count Decreased (Investigations) | 62 | 50
Lymphocyte Count Decreased (Investigations) | 31 | 30
Alanine Amino Transferase Increased (Investigations) | 23 | 28
Weight decreased (Investigations) | 20 | 19
Aspartate Amino Transferase Increased (Investigations) | 18 | 27
Blood Bilirubin Increased (Investigations) | 17 | 12
Electrocardiogram QT prolonged (Investigations) | 17 | 11
GGT increased (Investigations) | 9 | 7
Blood LDH Increased (Investigations) | 8 | 5
EKG T wave abnormal (Investigations) | 8 | 2
Neutrophil Count Increased (Investigations) | 6 | 7
Blood Creatinine Increased (Investigations) | 5 | 9
Anemia (Blood and lymphatic system disorders) | 91 | 80
Neutropenia (Blood and lymphatic system disorders) | 28 | 25
Febrile Neutropenia (Blood and lymphatic system disorders) | 20 | 21
Leucopenia (Blood and lymphatic system disorders) | 15 | 22
Thrombocitopenia (Blood and lymphatic system disorders) | 14 | 17
Nausea (Gastrointestinal disorders) | 51 | 39
Vomiting (Gastrointestinal disorders) | 27 | 20
Constipation (Gastrointestinal disorders) | 26 | 30
Diarrhea (Gastrointestinal disorders) | 23 | 20
Stomatitis (Gastrointestinal disorders) | 17 | 12
Abdominal Pain (Gastrointestinal disorders) | 16 | 8
Abdominal Distension (Gastrointestinal disorders) | 7 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 7
Hypokalemia (Metabolism and nutrition disorders) | 23 | 34
Hyponatremia (Metabolism and nutrition disorders) | 23 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 14
Decreased Apetite (Metabolism and nutrition disorders) | 17 | 11
Hypokalcemia (Metabolism and nutrition disorders) | 11 | 15
Hyperuricemia (Metabolism and nutrition disorders) | 10 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 3
Pyrexia (General disorders) | 34 | 30
Fatigue (General disorders) | 22 | 21
Malaise (General disorders) | 18 | 15
Edema Peripheral (General disorders) | 13 | 17
Chills (General disorders) | 6 | 10
Non-Cardiac Chest Pain (General disorders) | 2 | 12
Peripheral Neuropathy (Nervous system disorders) | 19 | 12
Hypoaesthesia (Nervous system disorders) | 14 | 12
Dizziness (Nervous system disorders) | 13 | 18
Headache (Nervous system disorders) | 13 | 11
URTI (Infections and infestations) | 15 | 18
Pneumonia (Infections and infestations) | 12 | 11
Lung Infection (Infections and infestations) | 8 | 12
UTI (Infections and infestations) | 7 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 11
ILD (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 43
Infusion Related Reactions (Injury, poisoning and procedural complications) | 28 | 28
Sinus Tachycardia (Cardiac disorders) | 14 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 | 5
Hypertension (Vascular disorders) | 7 | 11
Hypotension (Vascular disorders) | 7 | 4
Chromaturia (Renal and urinary disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 16 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03263026/Prot_SAP_000.pdf